CLINICAL TRIAL: NCT02792257
Title: Pilot Trial of Dronabinol Adjunctive Treatment of Agitation in Alzheimer's Disease
Brief Title: Trial of Dronabinol Adjunctive Treatment of Agitation in Alzheimer's Disease
Acronym: THC-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Mclean Hospital (Other); Miami Jewish Health (Unknown); National Institute on Aging (NIA) (NIH); Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00052955; R01AG050515 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; Dementia; Cannabinoids; Agitation; Neuropsychiatric Symptoms
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychomotor Agitation | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dronabinol (Experimental): Study medication will be administered twice daily. Capsules of dronabinol will contain 2.5 mg per dose (5mg daily) during Week 1, then increase to 5 mg per dose (10mg daily) for Weeks 2 and 3.
  Interventions: Drug: Dronabinol (Marinol®)
- Placebo (Placebo Comparator): Placebo medication will be administered twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol (Marinol®) — 5mg - 10mg daily dose
  Arms: Dronabinol
Drug: Placebo — Daily dose
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is the most prevalent neurodegenerative disease of aging. Neuropsychiatric symptoms (NPS) in AD are a major cause of burden to patients, caregivers, and society and are near-universal at some point in the AD course. One of the most troubling of these symptoms is agitation (Agit-AD), typified by a variety of problem behaviors including combativeness, yelling, pacing, lack of cooperation with care, insomnia, and restlessness. There is a great need for better interventions that target Agit-AD, a major source of patient disability as well as caregiver burden and stress, particularly in the case of moderate to severe agitation. This pilot trial could open the door to "re-purposing" Dronabinol (Marinol®) as a novel and safe treatment for Agit-AD with significant public health impact.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most prevalent neurodegenerative disease of aging, affecting an estimated 5.2 million Americans and predicted to increase to 13.8 million by 2050. AD affects both cognition and emotion. Neuropsychiatric symptoms (NPS) in AD are a major cause of burden to patients, caregivers, and society and are near-universal at some point in the AD course with > 97% of AD patients having at least one symptom reported on the Neuropsychiatric Inventory (NPI).

One of the most troubling of these symptoms is agitation (Agit-AD), typified by a variety of problem behaviors including combativeness, yelling, pacing, lack of cooperation with care, insomnia, and restlessness. In community-based samples, Agit-AD is common. Agit-AD is associated with greater caregiver burden and shorter time to institutionalization, and there is a particularly acute need for interventions for severe Agit-AD in advanced dementia.

While there are currently no FDA approved medications for Agit-AD, psychotropic medications are widely prescribed "off-label" to treat Agit-AD. The most commonly used classes of medications prescribed for "off-label" treatment are antipsychotics and antidepressants. The evidence to date for efficacy remains mixed. Antipsychotics appear to have some degree of efficacy, but the effects are not highly replicable and it's use is associated with increased mortality in elderly patients with dementia. Antidepressants (particularly selective serotonin reuptake inhibitors, (SSRI)s) appear to have fewer and less severe adverse effects compared to antipsychotics, as well as no known mortality risks, but are not without limitation. Therefore, exploration of alternative treatments for Agit-AD, particularly severe cases, is timely and warranted.

Dronabinol (Marinol®) is FDA-approved for the treatment of anorexia/weight loss in AIDS and for nausea/emesis associated with chemotherapy, which is now being used off-label for Agit-AD. Dronabinol is a synthetic oral formulation of delta-9-tetrahydrocannabinol (THC), a psychoactive constituent of the cannabis plant that acts as a partial agonist at the Type 1 (CB1) and Type 2 (CB2) endocannabinoid receptors. This pharmacology is appropriate for targeting Agit-AD because CB1 receptor agonism can produce anxiolytic and antidepressant effects and CB2 receptor agonism can be anti-inflammatory.

The mechanism by which dronabinol exerts its effects on agitation and aggression in patients with dementia may occur through its action at the CB1 and/or the CB2 receptor. Agonists at the CB1 receptor in the brain improve anxiety and depression in humans as well as animal models. Dronabinol is an effective agonist at the CB1 receptor, which is generally specific to neurons and localized predominantly on the presynaptic terminal where it inhibits glutamatergic, dopaminergic and other neurotransmitter release. The CB1 receptor effects has been observed to mediate the observed anxiolytic and antidepressant effects of THC. Dronabinol is also an agonist at CB2, a potent anti-inflammatory receptor localized on activated microglia. Patients with AD have increased central and peripheral inflammation, likely as a result of the accumulation of beta-amyloid. Increased inflammation may have a number of behavioral effects that could drive the agitation and aggression in dementia patients. Dronabinol's effects at the CB2 receptor therefore could also produce changes in behavior in AD patients by reducing inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Dementia due to AD
2. Presence of Agit-AD as defined by the provisional criteria from the International Psychogeriatric Association (IPA). The definition requires the presence of cognitive impairment, evidence of emotional distress, one of three observable types of behavior (excessive motor activity, verbal aggression, physical aggression), requires that the behavior cause excess disability, and notes that the behaviors cannot be solely attributable to another disorder such as psychiatric illness, medical illness, or effects of substance use.
3. Clinically significant severity of agitation defined by NPI-C Agitation or NPI-C Aggression > 4.
4. Able to give informed consent, or deemed to lack such capacity by clinical team and legally authorized representative consents.
5. Must be fluent in English and/or Spanish (includes reading, writing, and speech)
6. Must be admitted to clinical sites associated with McLean Hospital, Johns Hopkins University, and Miami Jewish Health Services as an inpatient/long term care resident during the study duration (3 weeks) OR be able to travel to these locations to enroll as an outpatient.
7. Must be 60-95 years old
8. Must begin enrollment in study within one week of being determined eligible

Exclusion Criteria:

1. Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease, which might confound assessment of safety outcomes.
2. Seizure disorder
3. Baseline delirium as determined by Confusion Assessment Method (CAM) and Diagnostic and Statistical Manual of Mental Disorders (DSM) -5 criteria
4. Current use of lithium
5. Inability to swallow a pill

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rosenberg, Principal Investigator — Johns Hopkins University; Brent Forester, Principal Investigator — Tufts Medical Center
Locations (5):
- United States (5):
  - Miami Jewish Health, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - North Shore Medical Center, Salem, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of study completion
Access Criteria: Investigators will send a proposal to the principal investigators (Drs. Rosenberg and Forester) who will decide if the proposal is satisfactory and if so, send the information listed above.

REFERENCES:
- [Derived] Rosenberg PB, Amjad H, Burhanullah H, Nowrangi M, Vandrey R, Pierre MJ, Outen JD, Schultz M, Marano C, Agronin M, Wilkins JM, Harper D, Laffaye T, Reardon E, Turner K, Ozonsi R, Drury M, Nguyen A, Hasoglu T, Cromwell J, Leoutsakos JM, Forester BP. A Randomized Controlled Trial of the Safety and Efficacy of Dronabinol for Agitation in Alzheimer's Disease. Am J Geriatr Psychiatry. 2026 Feb;34(2):167-179. doi: 10.1016/j.jagp.2025.10.011. Epub 2025 Nov 10. PMID 41350162
- [Derived] Cohen LM, Ash E, Outen JD, Vandrey R, Amjad H, Agronin M, Burhanullah MH, Walsh P, Wilkins JM, Leoutsakos JM, Nowrangi MA, Harper D, Rosenberg PB, Forester BP. Study rationale and baseline data for pilot trial of dronabinol adjunctive treatment of agitation in Alzheimer's dementia (THC-AD). Int Psychogeriatr. 2024 Dec;36(12):1245-1250. doi: 10.1017/S1041610221001150. Epub 2021 Oct 11. PMID 34629131
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852
- [Derived] Solomon HV, Greenstein AP, DeLisi LE. Cannabis Use in Older Adults: A Perspective. Harv Rev Psychiatry. 2021 May-Jun 01;29(3):225-233. doi: 10.1097/HRP.0000000000000289. PMID 33660625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 84 enrolled participants at 5 clinical research sites. Most of the recruitment was at three sites (Johns Hopkins, McLean, and Miami).
Pre-assignment Details: 84 subjects signed consents to be screened for eligibility. 9 participants signed consents but did not meet the eligibility criteria to start the study (screen failures). 75 subjects were randomized to treatment groups in the study.
Period: Overall Study
Arm/Group | Dronabinol | Placebo
Started | 37 | 38
Completed | 32 | 31
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 3 | 4
Not completed — Allergy | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Excessive Agitation | 0 | 1
Not completed — Not Feeling Well | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol | Placebo | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean Age | 79.1 (7.3) | 77.9 (7.7) | 78.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 33 | 34 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 35 | 32 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Mean (Standard Deviation); unit: years] | 14.1 (2.9) | 13.6 (3.6) | 13.8 (3.2)
Current Antidepressant [Count of Participants; unit: Participants]
  Yes | 7 | 25 | 32
  No | 30 | 13 | 43
Current Antipsychotic [Count of Participants; unit: Participants]
  Yes | 20 | 18 | 38
  No | 17 | 20 | 37
NPI-C Agitation/Aggression [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory Clinician Rating Scale Agitation and Aggression section (NPI-C AA) is used for assessing agitation and aggression in those with dementia. The minimum score is 0 and the maximum in 63, with a higher score indicating a worse outcome and meaning more agitation.
  units on a scale | 21.9 (9.7) | 19.0 (11.2) | 20.4 (10.5)
NPI-C Sleep [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory Clinician Rating Scale- Sleep section (NPI-C Sleep) is to assess sleep symptoms and sleep disturbances in those with dementia. The minimum score is 0 and the max is 24. A higher number indicates a worse outcome (more sleep disturbance).
  units on a scale | 3.3 (5.1) | 3.6 (4.9) | 3.5 (5.0)
NPI-C Disinhibition [Mean (Standard Deviation); unit: units on a scale] — The The Neuropsychiatric Inventory Clinician Rating Scale- Disinhibition (NPI-C Disinhibition) is a subset of questions used to assess disinhibition in those with dementia. The minimum score is 0 and the maximum is 48. A higher score indicates a worse outcome or more disinhibition.
  units on a scale | 7.4 (7.3) | 5.8 (7.0) | 6.6 (7.1)
NPI-C Irritability [Mean (Standard Deviation); unit: units on a scale] — The NPI-C (Neuropsychiatric Inventory Clinician Rating Scale)- Irritability is used to assess irritability symptoms in dementia. The minimum is 0 and the max is 36. A higher number indicates more irritability.
  units on a scale | 10.3 (7.6) | 10.3 (9.9) | 10.3 (8.8)
Activities of Daily Living (ADL) Checklist [Mean (Standard Deviation); unit: units on a scale] — ADL (Activities of Daily Living) is a checklist that is used to determine how well you can do activities of daily living. The minimum is 0 (meaning very dependent) and the maximum is 78 (meaning very independent). A higher score is a better outcome meaning the person is more independent.
  units on a scale | 25.4 (20.3) | 21.1 (19.2) | 23.2 (19.8)
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The MMSE (Mini Mental State Exam) is used to assess cognitive function, particularly in individuals with cognitive impairment. The minimum is 0 and the maximum is 30. A higher score means the patient is able to function better.
  units on a scale | 9.1 (7.8) | 8.2 (5.7) | 8.6 (6.8)
Severe Impairment Battery (SIB) [Mean (Standard Deviation); unit: units on a scale] — The SIB 8 (severe impairment battery) is an 8 item version designed to assess cognitive function in patients with advanced dementia. The minimum score is 0 and the maximum is 16. a higher score indicates a worse outcome or more severe cognitive impairment.
  units on a scale | 11.9 (7.4) | 12.6 (6.3) | 12.3 (6.8)
Cohen Mansfield Agitation Inventory (CMAI) [Mean (Standard Deviation); unit: units on a scale] — The Cohen-Mansfield Agitation Inventory (CMAI) is used to assess agitation. The minimum is 14 and the maximum is 70. A higher number indicates a worse outcome, meaning there is more agitation.
  units on a scale | 30.5 (7.9) | 28.9 (9.1) | 29.7 (8.5)
NPI-C Total [Mean (Standard Deviation); unit: units on a scale] — This is the The Neuropsychiatric Inventory Clinician Rating Scale and is used to assess cognitive impairment in those with dementia with a min score of 0 and a max of 426. A higher score indicates a worse outcome or more severe impairment.
  units on a scale | 76.7 (34.2) | 76.4 (48.6) | 76.5 (41.8)
NPI-C Caregiver Distress [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory Clinician Rating Scale for caregiver distress (NPI-C Caregiver Distress) incorporates a measure of caregiver distress for people caring for those with dementia. The minimum score is 0 and the maximum score is 710, and a higher score indicates more caregiver distress.
  units on a scale | 89.8 (57.4) | 81.2 (72.9) | 85.4 (65.4)
Pittsburgh Agitation Scale (PAS) [Mean (Standard Deviation); unit: units on a scale] — The PAS (Pittsburgh Agitation Scale) assesses agitation in dementia patients with a minimum score of 0 and a maximum score of 16. A higher score means indicates the presence of more severe agitation.
  units on a scale | 7.1 (4.1) | 5.6 (4.2) | 6.3 (4.2)
Confusion Assessment Method (CAM) [Count of Participants; unit: Participants] — Confusion Assessment Method (CAM) is a standardized tool used to identify and diagnose delirium, a state of acute confusion.
  Participants
    0, Alert | 32 | 36 | 68
    1, Vigilant | 2 | 1 | 3
    1, Lethargic | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Agitation as Measured by the Pittsburgh Agitation Scale
Description: The Pittsburgh Agitation Scale (PAS) is a tool used to assess the severity of agitation in patients, particularly with dementia. The minimum score is 0 and the maximum score is 16. A higher number means a worse outcome, meaning more agitation.
Time Frame: Up to 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 37 | 38
score on a scale
  Week 0 | 7.14 (4.12) | 5.55 (4.18)
  Week 1 | 5.69 (4.36) | 4.97 (3.81)
  Week 2 | 5.73 (4.67) | 5.22 (4.24)
  Week 3 | 4 (3.52) | 5.13 (4.44)
Statistical Analysis 1: Comparison: Dronabinol vs Placebo; Efficacy is assessed by fitting a longitudinal linear GEE model with the co primary outcomes and with time, treatment arm, and their interaction. Analyses are adjusted for site and for use of antidepressants and antipsychotics at baseline. The treatment by week interaction is the coefficient of interest and represents the difference in change in outcome per week between the two arms; Test type: Superiority; p = .015, Regression, Linear; Difference in slopes = -0.74, 95% CI 2-sided [-1.328 to -0.152], Standard Error of Mean 0.3 — standard error NOT standard error of the mean

2. Primary Outcome: Symptoms of Agitation as Measured by the Neuropsychiatric Inventory, Clinician Version
Description: The Neuropsychiatric Inventory Clinician Version (NPI-C) is an assessment tool used to evaluate neuropsychiatric symptoms in patients, particularly those with dementia. The minimum score is 0 and the max is 426. Higher scores indicate worse outcomes, meaning more agitation.
Time Frame: Up to 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 37 | 38
score on a scale
  Week 0 | 76.68 (34.19) | 76.37 (48.62)
  Week 1 | 59 (37.95) | 56.54 (48.07)
  Week 2 | 55.56 (41.73) | 56.59 (47.38)
  Week 3 | 52.38 (38.21) | 51.06 (46.9)
Statistical Analysis 1: Comparison: Dronabinol vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .094, Regression, Linear; Difference in slopes = -1.26, 95% CI 2-sided [-2.73 to 0.21], Standard Error of Mean 0.75 — standard error not standard error of the mean

3. Secondary Outcome: Number of Participants With Adverse Events in Dronabinol Treatment as Compared to Placebo
Description: All Adverse Events (AE) s occurring after randomization and during the 3-week treatment period, regardless of adherence to study treatment, will be recorded at all contacts.
Time Frame: Up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 37 | 38
Participants
  0 AEs | 16 | 18
  1 AEs | 10 | 11
  2 AE | 6 | 5
  3 AE | 3 | 1
  4 AE | 1 | 2
  5 AE | 0 | 1
  8 AE | 1 | 0
Statistical Analysis 1: Comparison: Dronabinol vs Placebo; Test type: Superiority; p = .57, Regression, Logistic; The original analytic plan called for a logistic regression of ever/never SAE as a function of treatment assignment; Incident rate ratio = 1.14, 95% CI 2-sided [0.73 to 1.79], Standard Error of Mean 0.26 — not standard error of the mean just standard error

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Description: Serious adverse events were defined per FDA guidelines and reported in a timely manner.
Arm/Group | Dronabinol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/38
Other Adverse Events (participants affected / at risk) | 21/37 | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=37) | Placebo (N=38)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0) — participant experienced this twice
Humeral Fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=37) | Placebo (N=38)
Delirium (Psychiatric disorders) | 1 (1) | 2 (3)
Fall (General disorders) | 3 (4) | 5 (6)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 0 (0)
Urine Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Edema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 0 (0)
Neuroleptic Malignant Syndrome (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Prostatitis (Infections and infestations) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1) | 1 (1)
Pressure Ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Required Pain Management (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Appetite, Decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Appetite, Increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 5 (7)
Agitation (Psychiatric disorders) | 2 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ingrown Toenail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02792257/Prot_SAP_000.pdf